CLINICAL TRIAL: NCT01144039
Title: Glutamate Infusion in Hypertrophied Ventricle After Aortic Valve Replacement - a Randomized Trial
Brief Title: Glutamate and Diastolic Function in Patients Undergoing Aortic Valve Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: VI_echo_01_2006
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2008-09

CONDITIONS: Hypertrophy, Left Ventricular; Aortic Stenosis; Myocardial Ischemia; Cardiopulmonary Bypass
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Aortic Valve Stenosis; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: LG-group
Drug: HG-group
Drug: Placebo-group

SUMMARY:
Purpose: The effect of intravenous glutamate infusion on myocardial diastolic function and overall hemodynamics were studied in patients undergoing elective aortic valve replacement with severe aortic stenosis and associated left ventricular hypertrophy .

Methods: 25 patients will be included in this double-blind randomized placebo-controlled study. Glutamate was administered intravenously immediately after aortic cross-clamp release. The patients receive either a low dose of 30mg kg-1 h-1 (LG-group) or high dose of 60 mg kg-1 h-1 (HG-group) or placebo (P-group) at a rate of 3.3ml kg-1h-1 for 2h. Transesophageal echocardiography (TEE) is used to measure diastolic and systolic ventricular function before sternotomy (T0), and 2h (T2), 3h (T3) and 6h (T4) after release of cross clamp. Additionally routine hemodynamic parameters are measured intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* severe aortic stenosis
* left ventricular hypertrophy of more than 10mm IVS thickness
* normal ejection fraction
* SR

Exclusion Criteria:

* moderately or severely reduced systolic left ventricular function (ejection fraction <30%)
* atrial fibrillation or flutter
* intolerance to glutamate.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-02; Primary Completion 2007-11 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
flow propagational velocity
Isovolumic relaxation time
E-velocity
A-velocity
E/A ratio

SECONDARY OUTCOMES:
ejection fraction
cardiac output
mitral ring motion

CONTACTS AND LOCATIONS:
Locations (1):
- Clin. Dept. of Cardiothoracic and Vascular Anaesthesia & Intensive Medicine, Medical University of Vienna, Vienna General Hospital, Vienna, Vienna, Austria